CLINICAL TRIAL: NCT00784017
Title: Comparative Efficacy and Safety of Two Asparaginase Preparations in Children With Previously Untreated Acute Lymphoblastic Leukaemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MC-ASP.5/ALL; EudraCT number 2006-003180-31
Record Dates: First submitted 2008-10-31; First posted 2008-11-03 (Estimated); Last update posted 2013-02-27 (Estimated); Status verified 2013-02

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: Children with previously untreated acute lymphoblastic leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Asparaginase; asparaginase erwinia chrysanthemi recombinant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- asparaginase medac (Active Comparator)
  Interventions: Drug: asparaginase
- recombinant asparaginase (Experimental)
  Interventions: Drug: recombinant asparaginase

INTERVENTIONS:
Drug: asparaginase — 5.000U /m²; IV; day 12, 15, 18, 21, 24, 27, 30, 33
  Arms: asparaginase medac
Drug: recombinant asparaginase — 5.000U /m²; IV; day 12, 15, 18, 21, 24, 27, 30, 33
  Arms: recombinant asparaginase

SUMMARY:
This multicentric phase III study is designed to assess the efficacy and safety of recombinant asparaginase (rASNase) in comparison to Asparaginase medac™ during treatment of children with de novo ALL

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated T-lineage or precursor B-lineage ALL
* Patients must have morphological proof of ALL and diagnosis must be made from bone marrow morphology with more than 25% blasts
* Written informed consent
* Treatment according to DCOG ALL 10 protocol

Exclusion Criteria:

* Mature B-lineage ALL
* Patients with secondary ALL
* Known allergy to any ASNase preparation
* General health status according to Karnofsky / Lansky score < 40%
* Pre-existing known coagulopathy (e.g. haemophilia)
* Pre-existing pancreatitis
* Liver insufficiency (Bilirubin > 50 µmol/L; SGOT/SGPT > 10 x ULN)
* Other current malignancies
* Pregnancy (planned or existent), breast feeding

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 199 (Actual)
Dates: Start 2008-10; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
To determine the rate of patients with complete asparagine (ASN) depletion in serum during induction treatment and to demonstrate non-inferiority of rASNase compared to Asparaginase medac™ with respect to this parameter | March 2012

SECONDARY OUTCOMES:
To assess the incidence of patients with hypersensitivity reactions to the first dose of ASNase in the post-induction treatment | March 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

REFERENCES:
- [Derived] van der Sluis IM, de Groot-Kruseman H, Te Loo M, Tissing WJE, van den Bos C, Kaspers GJL, Bierings M, Kollen WJW, Konig T, Pichlmeier U, Kuhnel HJ, Pieters R. Efficacy and safety of recombinant E. coli asparaginase in children with previously untreated acute lymphoblastic leukemia: A randomized multicenter study of the Dutch Childhood Oncology Group. Pediatr Blood Cancer. 2018 Aug;65(8):e27083. doi: 10.1002/pbc.27083. Epub 2018 May 4. PMID 29727043